CLINICAL TRIAL: NCT02839772
Title: A Randomised Controlled Trial to Evaluate the Effect of a New Skin Care Regimen on Skin Barrier Function in Those With Podoconiosis in Ethiopia
Brief Title: An RCT to Evaluate the Effect of a New Skin Care Regimen on SBF in Those With Podoconiosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Hull (Other)
Collaborators: Procter and Gamble (Industry)
Responsible Party: Principal Investigator, Jill Brooks, PhD student, University of Hull
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHull
Record Dates: First submitted 2016-07-12; First posted 2016-07-21 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2016-08

CONDITIONS: Non-filarial Elephantiasis
Keywords: podoconiosis; glycerine; RCT; SBF; TEWL; SC hydration
MeSH Terms: conditions — Elephantiasis | interventions — Glycerol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Current skin care regimen (Active Comparator): Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in 6 litres of water with added sodium hypochlorite (0.0125%), air dried, thin layer of petrolatum jelly applied and Whitfields ointment if required for any fungal infection.
  Interventions: Other: Current skin care regimen
- Current skin regimen plus 2% glycerine (Experimental): Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in 1 litre of water with added sodium hypochlorite (0.0125%) and 2% glycerine, air dried, thin layer of petrolatum jelly applied and Whitfields ointment if required for any fungal infection.
  Interventions: Other: Current skin care regimen plus 2% glycerine added to soaking water

INTERVENTIONS:
Other: Current skin care regimen plus 2% glycerine added to soaking water
  Other Names: glycerine
  Arms: Current skin regimen plus 2% glycerine
Other: Current skin care regimen
  Arms: Current skin care regimen

SUMMARY:
An RCT (n=193) in two podoconiosis clinics in Ethiopia to evaluate the effectiveness of a research based skin management regimen compared to the current regimen. The experimental group added 2% glycerine to the current skin care regimen and used 1 litre of water in the water soak compared to the 6 litres used in the current regimen.

DETAILED DESCRIPTION:
Background. Podoconiosis (non-filarial elephantiasis) affects some of the poorest people in 20 countries in the world. In Ethiopia least 3 million people are affected with 17 million at risk. Irritant minerals (smectite, mica and quartz) from volcanic soil and pathogens enter skin breaches in the feet causing inflammation, lymphoedema and hyperkeratosis. Podoconiosis is preventable and treatable but is not curable. Current treatment consists of educating those with disease on its causes, prevention and treatment. Treatment taught in the Action on Podoconiosis (APA) Clinics consists of a daily hygiene regimen of washing the feet/legs with soap, soaking the feet and legs in water with sodium hypochlorite (NaOCI) (0.0125%) added as a disinfectant, air drying and the application of a thin layer of petrolatum jelly. Whitfields ointment (benzoic acid and salicylic acid) is applied to any fungal infections. Wearing shoes is encouraged but this does not offer complete protection against the alkaline soil.

Although the current treatment skin care regimen is effective there is no robust evidence on optimal skin care regimens to improve skin barrier function in this disease.

Objective. To evaluate the effectiveness of a new, low-cost, evidence-based skin care intervention to improve SBF in the lower limbs of those with podoconiosis.

Method. A randomized control trial (RCT) was conducted over 3 months in two APA Clinics (n=193). Intervention was 2% glycerine (v/v) added to a reduced amount of soaking water (1 litre versus 6 litres). The control group received the current skin care regimen. The primary outcome measure was skin barrier function (SBF). This was determined by measures of trans-epidermal water loss (TEWL) and stratum corneum hydration (SCH) at four specific sites on the lower limbs.

ELIGIBILITY:
Inclusion Criteria:

* Patients in Ethiopia with a diagnosis of podoconiosis. That is those living above 1000 feet sea level with high rainfall, above 1,00mm annually with foot or lower leg oedema which had started in the feet, with sensation present in the feet and no hand involvement. The diagnosis was determined by the nurses at the outreach clinics.
* Patients who were able to understand instructions and give informed consent as determined by the nurses at the outreach clinics.
* Patients over 18 years of age.

Exclusion Criteria:

* Patients not diagnosed with podoconiosis as determined by nurses at the outreach clinics.
* Patients who were unable to understand instructions or give informed consent as determined by nurses at the outreach clinics.
* Patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Brooks, PhD student, Principal Investigator — University of Hull, UK; Steven J Ersser, PhD,, Study Director — University of Leeds, UK; Fiona C Cowdell, DProf,, Study Director — University of Hull, UK; Eric Gardiner, PhD,, Study Director — University of Hull, UK; Paul J Matts, PhD, Study Director — Procter and Gamble

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Current Skin Care Regimen: Legs/feet washed daily for 3 months with soapy water, soaked in 6 litres of water with added sodium hypochlorite (NaOCI) (0.0125%) and splashed up the lower legs with the hands for 30 mins, then air dried, a thin layer of petrolatum jelly applied. Whitfields ointment was applied if required to any areas of fungal infection.
- Current Skin Regimen Plus 2% Glycerine: Legs/feet washed daily for 3 months with soapy water, soaked in 1 litre of water with added sodium hypochlorite (NaOCI) (0.0125%) and splashed up the lower legs with the hands for 30 mins, then air dried, a thin layer of petrolatum jelly applied. Whitfields ointment was applied if required to any areas of fungal infection.
Period: Overall Study
Arm/Group | Current Skin Care Regimen | Current Skin Regimen Plus 2% Glycerine
Started | 97 (Stratification was used. Clinic A enrolled 94 participants and Clinic B 99 participants) | 96
Completed | 96 (1 participant in Clinic B did not return for the 3 months post- intervention data collection.) | 96
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Population: Clinic A. 47 with less severe/ moderate disease (stages 1,2,3) and 47 with severe disease (stages 4,5) Clinic B. 49 with less severe/ moderate disease and 50 with severe disease
Groups:
- Current Skin Care Regimen: Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in water with added sodium hypochlorite (NaOCI) (0.0125%), air dried, thin layer of petrolatum jelly applied. Whitfields ointment was applied if required to any areas of fungal infection.
- Current Skin Regimen Plus 2% Glycerine: Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in water with added sodium hypochlorite (NaOCI) (0.0125%) and 2% glycerine, air dried, thin layer of petrolatum jelly applied. Whitfields ointment was applied if required to any areas of fungal infection.
- Total: Total of all reporting groups
Arm/Group | Current Skin Care Regimen | Current Skin Regimen Plus 2% Glycerine | Total
Number analyzed (Participants) | 97 | 96 | 193
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 84 | 82 | 166
  >=65 years | 13 | 14 | 27
Gender [Count of Participants; unit: Participants]
  Female | 49 | 49 | 98
  Male | 48 | 47 | 95
Region of Enrollment [Number; unit: participants] — Data was collected from new patients attending two Action on Podoconiosis Clinics in south-central Ethiopia with similar graphical features. Clinical practice at both was the same.
  participants
    Ethiopia | 97 | 96 | 193
Severity of podoconioisis based on a staging systeme [Number; unit: participants] — There are 5 stages with 5 being the most severe stage of podoconiosis.
  participants
    Less severe/moderate disease | 47 | 46 | 93
    Severe disease | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in TEWL at Top of Outer Lower Legs
Description: Trans-epidermal water loss (TEWL) was measured with a Vapometer (non-invasive probe) on the outer lower leg 8 cms below the head of the fibula. TEWL is the water lost through the skin under non-sweating conditions. It is the major indicator of healthy skin. A reduction in TEWL indicates a positive effect on skin barrier function. It is generally recommended that differences or percentage changes are reported rather than absolute values.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data was missing from one male participant in the control group. One left leg in the control group and one right and one left leg in the experimental group was not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: g/m2/h
Units Other Than Participants: Legs
Groups:
- Control Group: Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in 6 litres of water with added sodium hypochlorite (NaOCI) (0.0125%), air dried, thin layer of petrolatum jelly applied. Whitfields ointment applied if required to any area of fungal infection.
- Experimental Group: Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in litre of water with added sodium hypochlorite (NaOCI) (0.0125%) and 2% glycerine and frequently splashed up legs, air dried, thin layer of petrolatum jelly applied. Whitfields ointment applied if required to any area of fungal infection.
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Legs) | 193 | 190
g/m2/h
  Right leg TEWL at 1st visit | 12.74 (4.73) | 13.43 (5.56)
  Left leg TEWL at 1st visit | 13.52 (5.61) | 13.27 (4.91)
  Right leg TEWL at 4th visit | 8.76 (2.63) | 7.06 (1.96)
  Left leg TEWL at 4th visit | 9.09 (2.63) | 7.53 (2.12)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function (SBF) in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in TEWL at the top of the outer lower legs by group from baseline after 3 months of interventions; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; t=5.341, df=89.347; Mean Difference (Final Values) = 1.581, 95% CI 2-sided [0.997 to 2.164], Standard Error of Mean 0.296

2. Primary Outcome: Change in TEWL at Mid-point Outer Lower Legs
Description: Trans-epidermal water loss (TEWL) was measured with a Vapometer (non- invasive probe) at a specific point on the outer lower leg. This was mid-way between the measurement site at the top of the outer leg and the site at the base of the outer lower leg. TEWL is the water lost through the skin under non-sweating conditions. It is the major indicator of healthy skin. A reduction in TEWL indicates a positive effect on skin barrier function. It is generally recommended that differences or percentage changes are reported rather than absolute values.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group. One left leg in the control group and one right and one left leg in the experimental group was not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: g/m2/h
Units Other Than Participants: Legs
Groups:
- Control Group: Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in water with added sodium hypochlorite (NaOCI) (0.0125%), air dried, thin layer of petrolatum jelly applied. Whitfields ointment applied if required to any area of fungal infection.
- Experimental Group: Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in 1 litre of water with added sodium hypochlorite (NaOCI) (0.0125%) and 2% glycerine and frequently splashed up legs, air dried, thin layer of petrolatum jelly applied. Whitfields ointment applied if required to any area of fungal infection.
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Legs) | 193 | 190
g/m2/h
  Right leg TEWL at 1st visit | 14.02 (5.12) | 14.57 (6.03)
  Left leg TEWL at 1st visit | 15.46 (6.07) | 14.55 (5.12)
  Right leg TEWL at 4th visit | 9.87 (2.86) | 8.22 (2.27)
  Left leg TEWL at 4th visit | 10.34 (3.27) | 8.61 (2.43)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in TEWL at the mid-point of the outer lower legs by group from baseline after 3 months of interventions; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; t=4.871, df=189.789; Mean Difference (Final Values) = 1.684, 95% CI 2-sided [1.002 to 2.367], Standard Error of Mean 0.346

3. Primary Outcome: Change in TEWL at Base of Outer Lower Legs
Description: Trans-epidermal water loss (TEWL) was measured with a Vapometer (non- invasive probe) at a specific point on the outer lower leg 8cms above the external malleolus. A reduction in TEWL indicates a positive effect on skin barrier function.It is generally recommended that differences or percentage changes are reported rather than absolute values.
  TEWL is the water lost through the skin under non-sweating conditions. It is the major indicator of healthy skin. A reduction in TEWL indicates a positive effect on skin barrier function. It is generally recommended that differences or percentage changes are reported rather than absolute values.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post-intervention data was missing from one male participant in control group.One left leg in the control group and one right and one left leg in the experimental group was not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: g/m2/h
Units Other Than Participants: Legs
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Legs) | 193 | 190
g/m2/h
  Right leg TEWL at 1st visit | 16.45 (6.13) | 16.80 (6.79)
  Left leg TEWL at 1st visit | 17.32 (5.46) | 17.02 (5.98)
  Right leg TEWL at 4th visit | 11.50 (3.35) | 9.30 (2.56)
  Left leg TEWL at 4th visit | 11.87 (3.59) | 9.88 (2.27)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in TEWL at the base of the outer lower legs by group from baseline after 3 months of interventions; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; t=5.111, df=189.620; Mean Difference (Final Values) = 1.970, 95% CI 2-sided [1.210 to 2.731], Standard Error of Mean 0.386

4. Primary Outcome: Change in TEWL at Top of Feet
Description: Trans-epidermal water loss (TEWL) was measured with a Vapometer (non- invasive probe) at a specific point on the top of the foot. A reduction in TEWL indicates a positive effect on skin barrier function.It is generally recommended that differences or percentage changes are reported rather than absolute values.
  TEWL is the water lost through the skin under non-sweating conditions. It is the major indicator of healthy skin. A reduction in TEWL indicates a positive effect on skin barrier function. It is generally recommended that differences or percentage changes are reported rather than absolute values.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in control group. One left foot leg in the control group and one right and one left foot in the experimental group was not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: g/m2/h
Units Other Than Participants: Feet
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Feet) | 193 | 190
g/m2/h
  Right foot 1st visit | 21.97 (5.46) | 22.88 (6.74)
  Left foot 1st visit | 23.01 (5.06) | 22.47 (6.79)
  Right foot 4th visit | 14.90 (4.36) | 13.15 (3.87)
  Left foot 4th visit | 15.38 (4.09) | 13.49 (3.77)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in TEWL at the top of the feet by group from baseline after 3 months of interventions; Test type: Superiority or Other; p = 0.002, Mixed Models Analysis; t=3.154, df=189.580; Mean Difference (Final Values) = 1.751, 95% CI 2-sided [0.656 to 2.846], Standard Error of Mean 0.390

5. Primary Outcome: Change in Stratum Corneum Hydration (SCH) at the Top of Outer Lower Legs
Description: Stratum corneum hydration was measured at a specific point at top of outer lower leg (8cms below the head of the fibula) with a MoistureMeter (non-invasive probe).This measures skin capacitance in arbitrary units. It is generally recommended that differences or percentage changes are reported rather than absolute values. Increases in stratum corneum hydration indicate a positive effect on skin barrier function.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in control group.One left leg in the control group and one right and one left leg in the experimental group was not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Units Other Than Participants: Legs
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Legs) | 193 | 190
Arbitrary units
  Right leg SCH 1st visit | 9.60 (3.96) | 9.05 (3.98)
  Left leg SCH 1st visit | 9.82 (4.54) | 9.25 (4.09)
  Right leg SCH 4th visit | 13.73 (3.59) | 16.24 (3.72)
  Left leg SCH 4th visit | 15.30 (11.19) | 16.10 (4.15)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in SCH at the top of the outer lower legs by group from baseline after 3 months of interventions; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; t=-4.236,df=165.310; Mean Difference (Final Values) = -2.075, 95% CI 2-sided [-3.042 to -1.1078], Standard Error of Mean 0.515

6. Primary Outcome: Change in Stratum Corneum Hydration (SCH) at Mid-point Outer Lower Leg.
Description: SCH was measured mid-way between the measurement site at the top of the outer leg and the site at the base of the outer lower leg. It was measured with a MoistureMeter (non-invasive probe).This measures skin capacitance in arbitrary units. It is generally recommended that differences or percentage changes are reported rather than absolute values. Increases in stratum corneum hydration indicate a positive effect on skin barrier function.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group.One left leg in the control group and one right and one left leg in the experimental group were not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Units Other Than Participants: Legs
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Legs) | 193 | 190
Arbitrary units
  Right leg SCH at 1st visit | 9.20 (3.29) | 8.86 (4.08)
  Left leg SCH at 1st visit | 9.39 (3.83) | 9.05 (3.78)
  Right leg SCH at 4th visit | 13.88 (2.78) | 15.90 (3.77)
  Left leg SCH at 4th visit | 14.56 (3.90) | 15.95 (3.19)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in SCH at the mid-point of the outer lower legs by group from baseline after 3 months of interventions; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; t=-3.549, df=180.923; Mean Difference (Final Values) = -1.658, 95% CI 2-sided [-2.581 to -0.736], Standard Error of Mean 0.467

7. Primary Outcome: Change in Stratum Corneum Hydration at Base of Outer Lower Leg
Description: Stratum corneum hydration was measured at the base of the outer lower leg 8 cms above the external malleolus. It was measured with a MoistureMeter (non-invasive probe).This measures skin capacitance in arbitrary units. It is generally recommended that differences or percentage changes are reported rather than absolute values. Increases in stratum corneum hydration indicate a positive effect on skin barrier function.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month data missing from one male participant in control group.One left leg in the control group and one right and one left leg in the experimental group were not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Units Other Than Participants: Legs
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Legs) | 193 | 190
Arbitrary units
  Right leg SCH 1st visit | 8.46 (3.95) | 8.56 (4.66)
  Left leg SCH at 1st visit | 8.26 (4.01) | 8.85 (4.36)
  Right leg SCH 4th visit | 14.25 (3.84) | 15.93 (3.80)
  Left leg SCH 4th visit | 14.47 (4.41) | 16.47 (3.40)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in SCH at the base of the outer lower legs by group from baseline after 3 months of interventions; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis; t=-3.471, df=186.308; Mean Difference (Final Values) = -1.641, 95% CI 2-sided [-2.574 to -0.708], Standard Error of Mean 0.473

8. Primary Outcome: Change in Stratum Corneum Hydration at Top of Feet
Description: Stratum corneum hydration measured at a specific point on the middle top of the foot with a MoistureMeter (non-invasive probe).This measures skin capacitance in arbitrary units. It is generally recommended that differences or percentage changes are reported rather than absolute values. Increases in stratum corneum hydration indicate a positive effect on skin barrier function.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group. One left foot in the control group and one left and one right foot in the experimental group were not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Units Other Than Participants: Feet
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Feet) | 193 | 190
Arbitrary units
  Right leg SCH at 1st visit | 8.48 (5.52) | 8.50 (6.30)
  Left leg SCH at 1st visit | 8.39 (5.97) | 8.87 (6.72)
  Right leg SCH at 4th visit | 15.31 (4.54) | 17.29 (4.59)
  Left leg SCH 4th visit | 15.14 (4.92) | 17.47 (4.90)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis compared the changes in SCH at the base of the top of the feet by group from baseline after 3 months of interventions; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; t=-3.565, df=186.739; Mean Difference (Final Values) = -2.041, 95% CI 2-sided [-3.168 to -0.911], Standard Error of Mean 0.572

9. Secondary Outcome: Stage of Podoconiosis in Each Leg of All Participants at Baseline and 4th Visit
Description: Podoconiosis Staging System (1-5) used with 5 the most severe stage. This staging system was specifically designed for those with podoconiosis. Legs with stages 1, 2 or 3 were categorised with mild/moderate disease and those with stages 4,5 with severe disease.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group. One leg in the control group and two legs in experimental group were not affected by podoconiosis. Data were pre-specified to be collected and analysed for all participants as a single group.
Measure: Number; unit: Legs/feet
Units Other Than Participants: Legs
Groups:
- Stage of Podoconiosis 1st Visit; Stage of Podoconiosis 4th Visit: The number of legs with each stage of podoconiosis (1-5) and those with no disease
Arm/Group | Stage of Podoconiosis 1st Visit | Stage of Podoconiosis 4th Visit
Number analyzed (Participants) | 193 | 192
Number analyzed (Legs) | 383 | 381
Legs/feet
  Right leg stage nil | 2 | 2
  Left legs stage nil | 1 | 1
  Right legs stage 1 | 22 | 56
  Left legs stage 1 | 20 | 49
  Right leg stage 2 | 63 | 50
  Left leg stage 2 | 66 | 53
  Right leg stage 3 | 19 | 64
  Left leg stage 3 | 17 | 68
  Right leg stage 4 | 72 | 29
  Left leg stage 4 | 75 | 21
  Right leg stage 5 | 15 | 0
  Left leg stage 5 | 14 | 0
  Right leg missing data | 0 | 1
  Left leg missing data | 0 | 1
Statistical Analysis 1: Comparison: Stage of Podoconiosis 1st Visit vs Stage of Podoconiosis 4th Visit; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis calculated the odds of the stage of podoconiosis by group being more severe at the 4th visit; Test type: Superiority or Other; p = 0.076, Generalized estimating equation analysis — A cumulative logistic link function was used; Wald Chi squared=3.138, df=1; Odds Ratio, log = 0.452, 95% CI 2-sided [-0.048 to 0.952], Standard Error of Mean 0.255

10. Secondary Outcome: Total Number of Trophic Skin Changes (Mossy Changes) All Participants at Baseline and 4th Visit
Description: Total number of observed trophic changes (mossy eruptions on the skin of the lower legs/feet characteristic of podoconiosis) in all participants by clinic nurse at baseline and at 4th visit. Trophic changes were either present or not present.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group.One leg in the control group and two legs in experimental group were not affected by podoconiosis. Data were pre-specified to be collected and analysed for all participants in a single group.
Measure: Number; unit: Trophic skin changes
Groups:
- Total Number of Trophic Skin Changes at Baseline: Trophic (mossy) skin changes on the lower legs/feet are a characteristic of podoconiosis. The total number of all participants with trophic changes in their lower legs/feet is reported.
- Total Number of Trophic Skin Changes at 4th Visit: Trophic (mossy) skin changes on the lower legs/feet are a characteristic of podoconiosis. The total number of all participants with trophic changes in their lower legs/feet is reported. A reduction in the number of legs/feet with mossy changes would denote an improvement in the condition.
Arm/Group | Total Number of Trophic Skin Changes at Baseline | Total Number of Trophic Skin Changes at 4th Visit
Number analyzed (Participants) | 193 | 192
Trophic skin changes | 312 | 237
Statistical Analysis 1: Comparison: Total Number of Trophic Skin Changes at Baseline vs Total Number of Trophic Skin Changes at 4th Visit; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis calculated the odds of mossy changes being present in the lower legs/feet by group at the 4th visit; Test type: Superiority or Other; p = 0.527, Generalized estimating equation analysis — A Bernouilli distribution with a logistic link function was used; Wald chi-square=0.410, df=1; Odds Ratio, log = -0.224, 95% CI 2-sided [-0.469 to 0.917]

11. Secondary Outcome: Total Number of All Participants With the Presence of a Bad Odour Emanating From Their Lower Limbs.
Description: Change in the presence of bad odour emanating from wounds on participant's lower legs/feet as determined by clinic nurse. Bad odour results in social stigma and impacts of quality of life.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group. One leg in the control group and two legs in experimental group were not affected by podoconiosis. Data were pre-specified to be collected and analysed for all participants in a single group.
Measure: Number; unit: Participants
Groups:
- Participants With Bad Odour From Legs/Feet at Baseline; Participants With Bad Odour From Legs/Feet at 4th Visit: Presence of a bad odour emanating from legs/feet of all participants as determined by clinic nurse.
Arm/Group | Participants With Bad Odour From Legs/Feet at Baseline | Participants With Bad Odour From Legs/Feet at 4th Visit
Number analyzed (Participants) | 193 | 192
Participants | 114 | 3
Statistical Analysis 1: Comparison: Participants With Bad Odour From Legs/Feet at Baseline vs Participants With Bad Odour From Legs/Feet at 4th Visit; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis calculated the odds of participants having a bad odour emanating from their lower legs/feet by group at the 4th visit. Bad odour results in a decease in quality of life; Test type: Superiority or Other; p = 0.031, Generalized estimating equation analysis — A Bernouilli distribution with a logistic link function was used; Wald chi-square=8.304, df=1; Odds Ratio, log = -1.29, 95% CI 2-sided [-2.161 to -0.411], Standard Error of Mean 0.446

12. Secondary Outcome: Number of Wounds on Lower Legs/Feet of Participants.
Description: Observation and count of number of wounds (all breaches of the stratum corneum including areas of fungal infection) on lower legs/feet by clinic nurse.
  Breaches in the skin and areas of fungal infection are more likely to occur in those with an impaired skin barrier function.A reduction in the number of wounds indicates an improvement in SBF.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group. One leg in the control group and two legs in experimental group were not affected by podoconiosis. Data was pre-specified to be analysed for all participants as a single group.
Measure: Number; unit: Wounds
Units Other Than Participants: Feet/legs
Groups:
- Number of Wounds at Baseline: The total number of wounds (skin breaches including areas of fungal infection) of all participants on all legs/feet at baseline.
- Number of Wounds 4th Visit: The total number of wounds (skin breaches including areas of fungal infection) of all participants on all legs/feet at 4th visit.
Arm/Group | Number of Wounds at Baseline | Number of Wounds 4th Visit
Number analyzed (Participants) | 193 | 192
Number analyzed (Feet/legs) | 383 | 381
Wounds | 962 | 29
Statistical Analysis 1: Comparison: Number of Wounds at Baseline vs Number of Wounds 4th Visit; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis calculated the odds of wounds being present on the lower legs/feet of participants by group at the 4th visit; Test type: Superiority or Other; p = 0.005, Generalized estimating equation analysis — A Poisson distribution with a logarithmic link function was used; Wald chi-square=7.745, df=1; Odds Ratio, log = 2.062, 95% CI 2-sided [0.610 to 3.514], Standard Error of Mean 0.741

13. Secondary Outcome: Change in Number of Work Days Lost in Previous Month Due to Adenolymphangitis (ADL)
Description: Verbal questioning of participants by clinic nurse or social worker as to number of work days lost due to severe leg pain (adenolymphangitis). Questioning was used as most participants were illiterate.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group.One leg in the control group and two legs in experimental group were not affected by podoconiosis.Data were pre-specified to be analysed for all participants as a single group.
Measure: Number; unit: Number of work days lost.
Groups:
- Number of Days Work Days Lost by All Participants Baseline; Number of Days Lost by All Participants at 4th Visit: Number of days work lost in previous month due to adeno-lymphangitis. Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in water with added sodium hypochlorite (NaOCI) (0.0125%) and 2% glycerine, air dried, thin layer of petrolatum jelly applied. Whitfields ointment applied if required to any area of fungal infection.
Arm/Group | Number of Days Work Days Lost by All Participants Baseline | Number of Days Lost by All Participants at 4th Visit
Number analyzed (Participants) | 193 | 192
Number of work days lost. | 868 | 9
Statistical Analysis 1: Comparison: Number of Days Work Days Lost by All Participants Baseline; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Statistical analysis calculated the odds by group of having had fewer work days lost in the previous month at the 4th visit due to ADL; Test type: Superiority or Other; p = 0.058, Generalized estimation equation — A Poisson distribution with a logarithmic link function was used; df=1; Group ratio estimate = 2.090, 0.058% CI 2-sided [-0.069 to 4.250], Standard Error of Mean 1.102 — Those in the experimental group were expected to have fewer work days lost due to ADL

14. Secondary Outcome: Correlation Between Number of Work Days Lost Due to Adenolymphangitis and Number of Wounds
Description: Statistical calculation of the correlation between the number of work days lost in the previous month due to leg pain (adenolymphangitis) and the number of wounds present on the lower leg/foot. Wounds on the lower legs/feet may produce a bad odour.
Time Frame: From baseline monthly for 3 months
Population: 3 month post intervention data missing from one male participant in the control group. One leg in the control group and two legs in experimental group were not affected by podoconiosis.Data were pre-specified to be collected and analysed for all participants in a single group.
Measure: Number; unit: Spearman's correlation coefficient
Groups:
- Correlation Between Number of Wounds and Days Lost Due to ADL: Correlation between nuumber of work days lost in previous month due to ADL and number of wounds (all skin breaches including areas of fungal infection)
Arm/Group | Correlation Between Number of Wounds and Days Lost Due to ADL
Number analyzed (Participants) | 193
Spearman's correlation coefficient
  Correlation at baseline | 0.252
  Correlation at 2nd visit | 0.306
  Correlation at 3rd visit | 0.291
  Correlation at 4th visit | 0.265
Statistical Analysis 1: Comparison: Correlation Between Number of Wounds and Days Lost Due to ADL; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen; Test type: Superiority or Other; p < 0.001, Spearman's correlation coefficient — The p value was < 0.001 at all time points; The correlation at the 1st visit was 0.252, at the 2nd 0.306, at the 3rd 0.291 and at the 4th 0.265

15. Secondary Outcome: Change in Largest Lower Leg Circumference
Description: Measured by clinic nurse in centimetres with a disposable tape measure at the point of largest circumference on the foot.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group.One left leg in the control group and one right and one left leg in the experimental group was not affected by podoconiosis so they were not included in the study.
Measure: Mean (Standard Deviation); unit: Centimetres
Units Other Than Participants: Legs
Groups:
- Experimental Group: Legs/feet washed daily for 3 months with soapy water, soak for 30 mins in water with added sodium hypochlorite (NaOCI) (0.0125%) and 2% glycerine, air dried, thin layer of petrolatum jelly applied. Whitfields ointment applied if required to any area of fungal infection.
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Legs) | 193 | 190
Centimetres | -3.86 (2.82) | -4.14 (1.74)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. A reduction in leg circumference indicates an improvement in the disease; Test type: Superiority or Other; p = 0.158, Mixed Models Analysis; df=185.386; Median Difference (Final Values) = 0.288, 95% CI 2-sided [-0.113 to 0.690], Standard Error of Mean 0.204

16. Secondary Outcome: Change in Largest Foot Circumference
Description: as for outcome 15
Time Frame: Change from baseline following 3 months of intervention
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Centimetres
Units Other Than Participants: Foot circumference
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
Number analyzed (Foot circumference) | 193 | 190
Centimetres | -2.34 (2.73) | -2.90 (1.93)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. A reduction in foot circumference indicates an improvement in the disease; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; df=169.916, t=3.550; Mean Difference (Final Values) = 0.575, 95% CI 2-sided [0.255 to 0.895], Standard Error of Mean 0.162

17. Secondary Outcome: Amharic Dermatology Life Quality Index (DLQI)
Description: The Amharic version of the DLQI has been validated for use in Ethiopia where Amharic is the official working language. The index is divided into 4 sections covering leisure, work and school, personal relationships and treatment. The maximum score of 30 indicates a high impact on quality of life. The lowest score zero. A reduction in the number indicates an improvement in quality of life. Participants were verbally questioned by the clinic nurse or social worker as most participants were illiterate.
Time Frame: Change from baseline following 3 months of intervention
Population: 3 month post intervention data missing from one male participant in the control group.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Experimental Group
Number analyzed (Participants) | 97 | 96
units on a scale
  DLQI at baseline | 21.61 (5.82) | 21.07 (7.49)
  DLQI 4th visit | 4.12 (4.29) | 3.94 (3.82)
Statistical Analysis 1: Comparison: Control Group vs Experimental Group; The null hypothesis was that an evidence-based skin care intervention with added glycerine does not improve skin barrier function in the legs/feet or enhance the disease related quality of life of Ethiopian people with podoconiosis when compared to the control group using the current skin care regimen. Podoconiosis has a large effect on a person's quality of life. abnormal looking legs/feet, wounds and the related bad odour plus social isolation result in stigma and social isolation; Test type: Superiority or Other; p = 0.907, Mixed Models Analysis; t=-0.117, df=178.814; Mean Difference (Final Values) = -0.063, 95% CI 2-sided [-1.129 to 1.002], Standard Error of Mean 0.540

ADVERSE EVENTS:
Time Frame: 3 months
Description: Any adverse effects of the regimes on the skin of the lower legs/feet of all participants were noted by the clinic nurse.
Groups:
- Control Group: Legs/feet washed daily for 3 months with soapy water, soaked in 6 litres of water with added sodium hypochlorite (NaOCI) (0.0125%) and splashed up the lower legs with the hands for 30 mins, then air dried, a thin layer of petrolatum jelly applied. Whitfields ointment was applied if required to any areas of fungal infection.
- Experimental Group: Legs/feet washed daily for 3 months with soapy water, soaked in 1 litre of water with added sodium hypochlorite (NaOCI) (0.0125%) and splashed up the lower legs with the hands for 30 mins, then air dried, a thin layer of petrolatum jelly applied. Whitfields ointment was applied if required to any areas of fungal infection.
Arm/Group | Control Group | Experimental Group
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/96
Other Adverse Events (participants affected / at risk) | 0/97 | 0/96

LIMITATIONS AND CAVEATS:
The study was not blinded which would have strengthened credibility and limited bias.The groups were matched but factors such as diet and co-morbidities particularly relating to blood flow in the legs/feet were not collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No